CLINICAL TRIAL: NCT01320644
Title: A Study of Robotic Assisted Laparoscopic Sacral Colpopexy Using Alyte Mesh
Acronym: ALYTE
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Principal Investigator, Atlantic Health System
Other Study IDs: R10-06-005
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Mesh Erosion
Keywords: Uterine prolapse; vaginal prolapse; mesh erosion; urinary incontinence; bowel symptoms
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vaginal mesh placement

SUMMARY:
Robotic approach to sacral colpopexy is a relatively new procedure. The literature is scarce in regard to long term outcomes. This advanced procedure is offered at Morristown Memorial. THis protocol will review the one year outcome of patients who underwent this pocedure using a polypropylene mesh. These outcomes will incude anatomical and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Any patient receiving Robotic assisted laparoscopic sacral copopexy with polypropylene mesh
* >21 y.o

Exclusion Criteria:

* Graft material other than polypropylene mesh
* Enrollment in another study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be woman who underwent robotic assisted laparoscopic sacral colpopexy at Morristown Memorial Hospital for the correction of pelvic organ prolapse using synthetic polypropylene mesh
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Memorial Hospital, Morristown, New Jersey, United States